CLINICAL TRIAL: NCT00006007
Title: A Phase II Study of a Combination of MTA (LY231514) and Gemcitabine in Patients With Metastatic Breast Cancer
Brief Title: LY231514 Plus Gemcitabine in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-983253; NCI-2012-02348 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068015 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gemcitabine + pemetrexed (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8. pemetrexed disodium IV is administered over 10 minutes 90 minutes following gemcitabine on day 8. Treatment continues every 21 days for a minimum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients achieving a complete response receive 2 additional courses.
  Patients are followed every 3 months for 5 years.
  Interventions: Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining LY231514 plus gemcitabine in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the antitumor activity of pemetrexed disodium in combination with gemcitabine in the treatment of women with metastatic breast cancer who have received an anthracycline and a taxane in the adjuvant and/or metastatic setting and no more than 1 chemotherapy regimen for metastatic disease (unless these were a taxane and anthracycline).
* Determine the toxicity of this regimen in this patient population.
* Determine time to progression and overall survival of these patients receiving this regimen.

OUTLINE: Patients receive gemcitabine IV over 30 minutes on days 1 and 8. pemetrexed disodium IV is administered over 10 minutes 90 minutes following gemcitabine on day 8. Treatment continues every 21 days for a minimum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients achieving a complete response receive 2 additional courses.

Patients are followed every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer with clinical evidence of metastatic disease
* Bidimensionally measurable disease

  * If bisphosphonates used, must have measurable disease site other than bone
  * No bone only disease
* Must have received a prior anthracycline and taxane in the adjuvant and/or metastatic setting
* No clinically significant pericardial effusions, pleural effusions, or ascites unless they can be drained
* No active CNS metastases

  * Treated CNS metastasis that has ben stable for at least 8 weeks allowed
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 3 times ULN (5 times ULN if liver metastases)
* Albumin at least 3.0 g/dL

Renal:

* Creatinine clearance at least 45 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to take folic acid and cyanocobalamin (vitamin B12) supplements
* Body surface area less than 3 m^2
* No uncontrolled infection
* No chronic debilitating disease
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated noninvasive carcinomas

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* At least 4 weeks since prior genetic therapy
* No concurrent immunomodulating agents

Chemotherapy:

* See Disease Characteristics
* No more than 3 prior chemotherapy regimens including adjuvant therapy

  * No more than 1 prior chemotherapy regimen for metastatic disease unless these were a taxane and anthracycline
* At least 4 weeks since prior chemotherapy
* No prior gemcitabine and/or pemetrexed disodium
* No other concurrent cytostatic or cytotoxic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to greater than 25% of bone marrow
* No prior strontium chloride Sr 89
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major surgery

Other:

* No aspirin or nonsteroidal antiinflammatory agents 2 days before, the day of, and for 2 days after pemetrexed disodium administration (5 days before for long acting agents such as naproxen, piroxicam, diflunisal, or nabumetone)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2000-12; Primary Completion 2004-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
time to progression | Up to 5 years

SECONDARY OUTCOMES:
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex A. Adjei, MD, PhD, Study Chair — Mayo Clinic
Locations (24):
- United States (23):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Ma CX, Steen P, Rowland KM, Niedringhaus RD, Fitch TR, Kugler JW, Hillman DW, Perez EA, Ingle JN, Adjei AA. A phase II trial of a combination of pemetrexed and gemcitabine in patients with metastatic breast cancer: an NCCTG study. Ann Oncol. 2006 Feb;17(2):226-31. doi: 10.1093/annonc/mdj054. Epub 2005 Nov 22. PMID 16303865
- [Result] Ma CX, Steen P, Rowland KM, et al.: A phase II study of a combination of pemetrexed (Pem) and gemcitabine (Gem) in patients with metastatic breast cancer (MBC): an NCCTG study. [Abstract] J Clin Oncol 22 (Suppl 14): A-639, 36s, 2004.